CLINICAL TRIAL: NCT01955720
Title: Randomised, Double-blind, Placebo-controlled, Two-way Cross-over Phase Ib Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of BI 655075 and to Establish the Efficacy of BI 655075 in Reversal of Dabigatran Anticoagulant Activity in Volunteers
Brief Title: Safety, Tolerability, PK and PD of BI 655075 and Establishment of BI 655075 Dose(s) Effective to Reverse Prolongation of Blood Coagulation Time by Dabigatran
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1321.2; 2013-003616-52 (EudraCT Number: EudraCT)
Record Dates: First submitted 2013-09-30; First posted 2013-10-07 (Estimated); Results first posted 2016-02-11 (Estimated); Last update posted 2016-02-11 (Estimated); Status verified 2016-01

CONDITIONS: Hemorrhage
MeSH Terms: conditions — Hemorrhage | interventions — idarucizumab

ARMS (4):
- healthy subjects aged 45-64 (Experimental): Sequential Crossover to Placebo or BI 655075
  Interventions: Drug: BI 655075; Drug: Placebo
- healthy elderly subjects aged 65-80 year (Experimental): Sequential Crossover to Placebo or BI 655075
  Interventions: Drug: BI 655075; Drug: Placebo
- mild renal impairment aged 45-80 years (Experimental): Sequential Crossover to Placebo or BI 655075
  Interventions: Drug: BI 655075; Drug: Placebo
- mod renal impairment aged 45-80 years (Experimental): Sequential Crossover to Placebo or BI 655075
  Interventions: Drug: Placebo; Drug: BI 655075

INTERVENTIONS:
Drug: BI 655075
  Arms: mild renal impairment aged 45-80 years
Drug: BI 655075
  Arms: healthy subjects aged 45-64
Drug: Placebo
  Arms: mod renal impairment aged 45-80 years
Drug: BI 655075
  Arms: healthy elderly subjects aged 65-80 year
Drug: Placebo
  Arms: healthy subjects aged 45-64
Drug: Placebo
  Arms: healthy elderly subjects aged 65-80 year
Drug: Placebo
  Arms: mild renal impairment aged 45-80 years
Drug: BI 655075
  Arms: mod renal impairment aged 45-80 years

SUMMARY:
To investigate safety, tolerability, PK and PD of BI 655075 and to establish the BI 655075 dose(s) effective to reverse prolongation of blood coagulation time by dabigatran

ELIGIBILITY:
Inclusion criteria:

* Healthy midage male and female volunteers, age =45 and =64 years, BMI range: =18.5 and =29.9 kg/m2
* Healthy elderly male and female volunteers, age =65 and =80 years, BMI range: =18.5 and = 32 kg/m2
* Male and female volunteers with mild renal impairment (CLcrd 60-90 (mL/min)) in relatively good health, age =45 and =80 years, BMI range: =18.5 and =32 kg/m2 Moderate renal impaired (CLcrd =30 to <60 mL/min according Cockcroft&Gault formula in relatively good health, age =45 and =80 years, BMI range: =18.5 and =32 kg/m2

Exclusion criteria:

* Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance
* Any evidence of a clinically relevant concomitant disease (other than mild renal impairment in the respective group) A significant disease is defined as a disease which in the opinion of the investigator
* put the volunteer at risk because of participation in the study
* may influence the results of the study
* may influence the volunteer¿s ability to participate in the study
* is not in a stable condition Diabetic, hypercholesterolemia or hypertensive subjects can be entered in this trial if the disease is not significant according to these criteria
* Surgery of the gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts.
* Chronic or relevant acute infections
* History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2013-09; Primary Completion 2014-05 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1321.2.1 Boehringer Ingelheim Investigational Site, Antwerp, Belgium

REFERENCES:
- [Derived] Norris S, Ramael S, Ikushima I, Haazen W, Harada A, Moschetti V, Imazu S, Reilly PA, Lang B, Stangier J, Glund S. Evaluation of the immunogenicity of the dabigatran reversal agent idarucizumab during Phase I studies. Br J Clin Pharmacol. 2017 Aug;83(8):1815-1825. doi: 10.1111/bcp.13269. Epub 2017 Apr 6. PMID 28230262
- [Derived] Glund S, Stangier J, van Ryn J, Schmohl M, Moschetti V, Haazen W, De Smet M, Gansser D, Norris S, Lang B, Reilly P, Kreuzer J. Effect of Age and Renal Function on Idarucizumab Pharmacokinetics and Idarucizumab-Mediated Reversal of Dabigatran Anticoagulant Activity in a Randomized, Double-Blind, Crossover Phase Ib Study. Clin Pharmacokinet. 2017 Jan;56(1):41-54. doi: 10.1007/s40262-016-0417-0. PMID 27317414
- [Derived] Glund S, Stangier J, van Ryn J, Schmohl M, Moschetti V, Haazen W, De Smet M, Gansser D, Norris S, Lang B, Reilly P, Kreuzer J. Restarting Dabigatran Etexilate 24 h After Reversal With Idarucizumab and Redosing Idarucizumab in Healthy Volunteers. J Am Coll Cardiol. 2016 Apr 5;67(13):1654-1656. doi: 10.1016/j.jacc.2016.01.043. No abstract available. PMID 27150693

RESULTS

PARTICIPANT FLOW:
Groups:
- 5 Ida / Placebo: Subjects received dabigatran (DE) 220 mg plus idarucizumab (Ida) 5g followed by dabigatran 220 mg plus placebo 5g (high dose)
- Placebo / 5 Ida: Subjects received dabigatran (DE) 220 mg plus placebo 5g followed by dabigatran 220 mg plus Ida 5g (high dose)
- 2.5 Ida / Placebo: Subjects received dabigatran (DE) 220 mg plus Ida 2.5g followed by dabigatran 220 mg plus placebo 2.5g (medium dose)
- Placebo / 2.5 Ida: Subjects received dabigatran (DE) 220 mg plus placebo 2.5g followed by dabigatran 220 mg plus Ida 2.5g (medium dose)
- 1 Ida / Placebo: Subjects received dabigatran (DE) 220 mg plus Ida 1g followed by dabigatran 220 mg plus placebo 1g (low dose)
- Placebo / 1 Ida: Subjects received dabigatran (DE) 220 mg plus placebo 1g followed by dabigatran 220 mg plus Ida 1g (low dose)
Period: Overall Study
Arm/Group | 5 Ida / Placebo | Placebo / 5 Ida | 2.5 Ida / Placebo | Placebo / 2.5 Ida | 1 Ida / Placebo | Placebo / 1 Ida
Started | 13 | 13 | 3 | 3 | 7 | 7
Healthy Subjects Aged 45-64 | 3 | 3 | 3 | 3 | 0 | 0
Healthy Subjects Aged 65-80 | 4 | 4 | 0 | 0 | 4 | 4
Subjects With Mild Renal Impairment | 3 | 3 | 0 | 0 | 3 | 3
Subjects With Moderate Renal Impairment | 3 | 3 | 0 | 0 | 0 | 0
Completed | 13 | 13 | 3 | 3 | 7 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set
Groups:
- Total Subjects Group: The total subjects group contains the following sub-groups: high dose (5 g idarucizumab), healthy, aged 45-64 yrs: high dose (5 g idarucizumab), healthy elderly, aged 65-80 yrs: high dose (5 g idarucizumab), mild renal impairment (RI), aged 45-80 yrs: high dose (2.5 g + 2.5 g idarucizumab), with moderate RI, aged 45-80 yrs: medium dose (2.5 g idarucizumab), healthy, aged 45-64 yrs: low dose (1 g idarucizumab), healthy elderly, aged 65-80 yrs: low dose (1 g idarucizumab), with mild RI, aged 45-80 yrs.
Arm/Group | Total Subjects Group
Number analyzed (Participants) | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.8 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 27

OUTCOME MEASURES:

1. Primary Outcome: Reversal of Dabigatran-induced Prolongation of Blood Coagulation Time
Description: Percentage of subjects with at least one assay value from diluted thrombin time (dTT) or ecarin clotting time (ECT) reversed within 10min after completion of infusion. Reversal was defined as return to baseline, where the threshold for reversal to baseline was determined using PK/PD correlation between unbound sum dabigatran and the clotting parameters ECT and dTT. Measured at the end of the infusion and 10 min later.
Time Frame: End of last infusion and 10 minutes after completion of last infusion of BI 655075
Population: PD Set (PDS): The PDS included all subjects from the TS who had at least 1 evaluable predose and on-treatment coagulation test measurement value for at least 1 coagulation test and who did not have important protocol violation relevant to the evaluation of PD.
Measure: Number; unit: percentage of participants
Groups:
- Placebo: idarucizumab-matching placebo
- Idarucizumab (Ida): Idarucizumab (Ida).
Arm/Group | Placebo | Idarucizumab (Ida)
Number analyzed (Participants) | 46 | 46
percentage of participants
  at least one time point, dTT | 0.0 | 100.0
  both time points, dTT | 0.0 | 100.0
  at least one time point, ECT | 0.0 | 100.0
  both time points, ECT | 0.0 | 100.0

2. Primary Outcome: The Percentage of Subjects With Drug-related Adverse Events
Description: The percentage of subjects with possibly drug-related AEs (as defined by the investigator) during the treatment period.
Time Frame: From baseline up to the start of follow-up period (from Day 1 to Day 35)
Population: Treated Set (TS): All randomised subjects who received at least 1 dose of trial medication were included in the treated set.
Measure: Number; unit: percentage of participants
Groups:
- On Treatment Group: during the treatment period.
Arm/Group | On Treatment Group
Number analyzed (Participants) | 46
percentage of participants | 13.0

3. Secondary Outcome: AUC0-infinity (Area Under the Concentration-time Curve of Idarucizumab (Ida) in Plasma Over the Time Interval From 0 Extrapolated to Infinity)
Description: AUC0-infinity. PK/PD sampling time: (p=predose, D=day)
  1. single medium or high dose, healthy subjects(HS) mid-age (45-64 yrs): D4: 8:55p, 9:00,9:10,9:30,10:00,11:00,13:00,15:00,19:00,21:00,01:00; D5: 9:00p, 21:00. D6: 9:00.
  2. single low or high dose, HS elderly or mild renal impaired: D4: 8:55p, 9:00,9:10,9:30,10:00,11:00,13:00,15:00,19:00,21:00,01:00; D5: 9:00; D6: 9:00; D7: 9:00; additional sampling for renal impaired: D8: 9:00;D9: 9:00.
  3. high 2 doses, moderate renal impaired: D4: 8:55p, 9:00, 9:10,9:30,9:55p, 10:00,10:10,10:30,11:00, 13:00, 15:00, 19:00, 21:00, 01:00; D5: 9:00; D6: 9:00; D7: 9:00; additional sampling for renal impaired: D8:9:00; D9:9:00.
Time Frame: From Day 4 to Day 9 (details in description)
Population: Pharmacokinetic Set -Ida (PKS-Ida): included all treated subjects who have received at least 1 dose of idarucizumab and who provided data for at least 1 secondary or other PK endpoint in any treatment period, which was judged as evaluable for PK and was not affected by protocol violations relevant to the statistical evaluation of PK endpoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Groups:
- 220 mg/2.5 g HS 45-64 Yrs: HS mid-age (45-64 yrs) with dabigatran (DE) 220 mg/Ida 2.5g.
- 220 mg/2.5 g HS 45-64 Yrs Re-exposure: HS mid-age (45-64 yrs) with dabigatran (DE) 220 mg/Ida 2.5g and reexposured Ida in period 3
- 220 mg/5 g HS 45-64 Yrs: HS mid-age (45-64 yrs) with dabigatran (DE) 220 mg/Ida 5g.
- 220 mg/1 g HS 65-80 Yrs: HS elderly (65-80 yrs) with dabigatran (DE) 220 mg/Ida 1g.
- 220 mg/5 g HS 65-80 Yrs: HS elderly (65-80 yrs) with dabigatran (DE) 220 mg/Ida 5g.
- 150 mg/1 g Mild Renal Impairment (RI): Mild RI (creatinine clearance [CL] 60-90) with dabigatran (DE) 150 mg/Ida 1g
- 150 mg/5 g Mild RI (CL 60-90): Mild RI (CL 60-90) with dabigatran (DE) 150 mg/Ida 5g
- 150 mg /2*2.5 g Moderate RI (CL 30-60): Moderate RI (CL 30-60) with dabigatran (DE) 150 mg and were infused 2 doses of each Ida 2.5g, given 1 h apart.
Arm/Group | 220 mg/2.5 g HS 45-64 Yrs | 220 mg/2.5 g HS 45-64 Yrs Re-exposure | 220 mg/5 g HS 45-64 Yrs | 220 mg/1 g HS 65-80 Yrs | 220 mg/5 g HS 65-80 Yrs | 150 mg/1 g Mild Renal Impairment (RI) | 150 mg/5 g Mild RI (CL 60-90) | 150 mg /2*2.5 g Moderate RI (CL 30-60)
Number analyzed (Participants) | 6 | 6 | 6 | 8 | 8 | 6 | 6 | 6
nmol*h/L | 22200 (12.7) | 20600 (10.6) | 37000 (18.4) | 8560 (15.2) | 43900 (18.7) | 10700 (14.1) | 53100 (11.1) | 67900 (11.6)

4. Secondary Outcome: AUC2-12, ss (Area Under the Concentration-time Curve of Unbound Sum Dabigatran (DE) in Plasma at Steady State Over the Time Interval From 2 to 12h)
Description: PK/PD sampling time:(d=dose,D=Day,p=predose)
  1. single medium or high dose,healthy, mid-age (45-64 yrs): D4: 7:00p,8:55p,9:00,9:10,9:30,10:00,11:00,13:00,15:00,19:00,21:00, 01:00; D5:9:00p,11:00,21:00p; D6:9:00p, 21:00p; D7:9:00p, 11:00.
  2. single low or high dose,healthy elder or mild renal impaired: D4:7:00p,8:55p,9:00,9:10,9:30,10:00,11:00,13:00,15:00,19:00,21:00,01:00;D5:9:00;D6:9:00;D7:9:00; additional sampling for renal impaired: D8:9:00;D9:9:00.
  3. high 2 doses, moderate renal impaired: D4:7:00p,8:55p,9:00,9:10,9:30,9:55p,10:00,10:10,10:30,11:00,13:00,15:00,19:00,21:00,01:00;D5:9:00;D6:9:00; D7:9:00; additional sampling for renal impaired: D8:9:00;D9:9:00.
Time Frame: from 2h to12h of post DE dose at steady state (details in description)
Population: PKS-DE: The PKS-DE included all treated subjects who have received at least 1 dose of DE and who provided data for at least 1 secondary or further PK endpoint in any treatment period, which was judged as evaluable for PK and was not affected by (important) protocol violations relevant to the statistical evaluation of PK endpoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- 220 mg/2.5g HS 45-64 Years: Healthy subjects (HS) mid-age (45-64 yrs) with dabigatran (DE) 220 mg/Ida 2.5g.
- 220 mg/Plc. 2.5g HS 45-64 Years: Healthy subjects (HS) mid-age (45-64 yrs) with dabigatran (DE) 220 mg/ placebo(plc.) 2.5g.
- 220 mg/2.5g HS 45-64 Yrs Re-exposure: Healthy subjects (HS) mid-age (45-64 yrs) with dabigatran (DE) 220 mg/Ida 2.5g and reexposured Ida in period 3
- 220 mg/5g HS 45-64 Yrs: Healthy subjects (HS) mid-age (45-64 yrs) with dabigatran (DE) 220 mg/Ida 5g
- 220 mg/Plc. 5g HS 45-64 Yrs: Healthy subjects (HS) mid-age (45-64 yrs) with dabigatran (DE) 220 mg/plc. 5g.
- 220 mg/1g HS 65-80 Yrs: Healthy subjects (HS) elderly (65-80 yrs) with dabigatran (DE) 220 mg/Ida 1g.
- 220 mg/Plc. 1g HS 65-80 Yrs: Healthy subjects (HS) elderly (65-80 yrs) with dabigatran (DE) 220 mg/plc. 1g.
- 220 mg/5g HS 65-80 Yrs: Healthy subjects (HS) elderly (65-80 yrs) with dabigatran (DE) 220 mg/Ida 5g.
- 220 mg/Plc. 5g HS 65-80 Yrs: Healthy subjects (HS) elderly (65-80 yrs) with dabigatran (DE) 220 mg/plc. 5g.
- 150 mg/1g Mild RI (CL 60-90): Mild RI (CL 60-90) with dabigatran (DE) 150 mg/Ida 1g
- 150 mg/Plc. 1g Mild RI (CL 60-90): Mild RI (CL 60-90) with dabigatran (DE) 150 mg/plc. 1g
- 150 mg/5g Mild RI (CL 60-90): Mild RI (CL 60-90) with dabigatran (DE) 150 mg/Ida 5g
- 150 mg/Plc. 5g Mild RI (CL 60-90): Mild RI (CL 60-90) with dabigatran (DE) 150 mg/plc. 5g
- 150 mg /2*2.5g Moderate RI (CL 30-60): Moderate RI (CL 30-60) with dabigatran (DE) 150 mg and were infused as 2 doses of each Ida 2.5g, given 1 h apart.
- 150 mg /Plc. 2*2.5g Moderate RI (CL 30-60): Moderate RI (CL 30-60) with dabigatran (DE) 150 mg and were infused as 2 doses of each plc. 2.5g, given 1 h apart.
Arm/Group | 220 mg/2.5g HS 45-64 Years | 220 mg/Plc. 2.5g HS 45-64 Years | 220 mg/2.5g HS 45-64 Yrs Re-exposure | 220 mg/5g HS 45-64 Yrs | 220 mg/Plc. 5g HS 45-64 Yrs | 220 mg/1g HS 65-80 Yrs | 220 mg/Plc. 1g HS 65-80 Yrs | 220 mg/5g HS 65-80 Yrs | 220 mg/Plc. 5g HS 65-80 Yrs | 150 mg/1g Mild RI (CL 60-90) | 150 mg/Plc. 1g Mild RI (CL 60-90) | 150 mg/5g Mild RI (CL 60-90) | 150 mg/Plc. 5g Mild RI (CL 60-90) | 150 mg /2*2.5g Moderate RI (CL 30-60) | 150 mg /Plc. 2*2.5g Moderate RI (CL 30-60)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 8 | 8 | 8 | 8 | 6 | 6 | 6 | 6 | 6 | 6
ng*h/mL | 18.5 (75.7) | 924 (25.6) | 36.0 (125) | 10.6 (11.3) | 933 (39.2) | 284 (66.3) | 1220 (40.0) | 11.6 (23.8) | 1270 (32.8) | 100 (192) | 929 (56.0) | 10.0 (0.0828) | 876 (40.5) | 10.2 (3.95) | 1440 (32.3)

5. Secondary Outcome: Aet1-t2, ss (Amount of DE Eliminated in Urine From the Time Point t1 to Time Point t2)
Description: Urinary excretion of sum dabigatran from the time point t1 to t2 at steady state.
  PK Urine sampling time:
  Urine sampling relative to first DE administration: Planned times 72:00 - 73:55h, 73:55 - 80:00h, 80:00 - 86:00h, 86:00 - 98:00h, 98:00 - 122:00h, 122:00 - 146:00h; additional sampling for renal impaired: 146:00 - 170:00; 170:00 - 194:00h.
  Ae0-26,ss was not measured in Period 3 (re-exposure period). Ae0-74,ss was not measured in healthy subjects aged 45 to 64 years.
Time Frame: From 0 to 74h post of last DE dose (details in description)
Population: Pharmacokinetic Set - DE (PKS-DE): The PKS-DE included all treated subjects who have received at least 1 dose of DE and who provided data for at least 1 secondary or further PK endpoint in any treatment period, which was judged as evaluable for PK and was not affected by protocol violations relevant to the statistical evaluation of PK endpoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg
Groups:
- 220 mg/2.5g HS 45-64 Years: HS mid-age (45-64 yrs) with dabigatran (DE) 220 mg/Ida 2.5g.
- 220 mg/Plc. 2.5g HS 45-64 Years: HS mid-age (45-64 yrs) with dabigatran (DE) 220 mg/ placebo(plc.) 2.5g.
- 220 mg/2.5g HS 45-64 Yrs Re-exposure: HS mid-age (45-64 yrs) with dabigatran (DE) 220 mg/Ida 2.5g and reexposured Ida in period 3
- 220 mg/5g HS 45-64 Yrs: HS mid-age (45-64 yrs) with dabigatran (DE) 220 mg/Ida 5g.
- 220 mg/Plc. 5g HS 45-64 Yrs: HS mid-age (45-64 yrs) with dabigatran (DE) 220 mg/plc. 5g.
- 220 mg/1g HS 65-80 Yrs: HS elderly (65-80 yrs) with dabigatran (DE) 220 mg/Ida 1g.
- 220 mg/Plc. 1g HS 65-80 Yrs: HS elderly (65-80 yrs) with dabigatran (DE) 220 mg/plc. 1g.
- 220 mg/5g HS 65-80 Yrs: HS elderly (65-80 yrs) with dabigatran (DE) 220 mg/Ida 5g.
- 220 mg/Plc. 5g HS 65-80 Yrs: HS elderly (65-80 yrs) with dabigatran (DE) 220 mg/plc. 5g.
Arm/Group | 220 mg/2.5g HS 45-64 Years | 220 mg/Plc. 2.5g HS 45-64 Years | 220 mg/2.5g HS 45-64 Yrs Re-exposure | 220 mg/5g HS 45-64 Yrs | 220 mg/Plc. 5g HS 45-64 Yrs | 220 mg/1g HS 65-80 Yrs | 220 mg/Plc. 1g HS 65-80 Yrs | 220 mg/5g HS 65-80 Yrs | 220 mg/Plc. 5g HS 65-80 Yrs | 150 mg/1g Mild RI (CL 60-90) | 150 mg/Plc. 1g Mild RI (CL 60-90) | 150 mg/5g Mild RI (CL 60-90) | 150 mg/Plc. 5g Mild RI (CL 60-90) | 150 mg /2*2.5g Moderate RI (CL 30-60) | 150 mg /Plc. 2*2.5g Moderate RI (CL 30-60)
Number analyzed (Participants) | 6 | 6 | 0 | 6 | 6 | 8 | 8 | 8 | 8 | 6 | 6 | 6 | 6 | 6 | 6
μg
  Ae0-26,ss(N=6,6,0,6,6,8,8,8,8,6,6,6,6,6,6) | 6080 (26.5) | 7460 (21.0) |  | 7560 (47.2) | 7790 (43.9) | 8490 (29.4) | 8870 (41.8) | 7460 (39.6) | 10600 (21.9) | 5800 (39.0) | 6040 (44.7) | 4020 (58.3) | 6280 (38.4) | 4760 (26.7) | 8880 (29.8)
  Ae0-74,ss(N=0,0,0,0,0,8,8,8,8,6,6,6,6,6,6) | NA (NA) — not measured in healthy subjects aged 45 to 64 years. | NA (NA) — not measured in healthy subjects aged 45 to 64 years. |  | NA (NA) — not measured in healthy subjects aged 45 to 64 years. | NA (NA) — not measured in healthy subjects aged 45 to 64 years. | 10700 (22.0) | 10300 (40.8) | 13900 (26.1) | 12800 (20.6) | 7760 (38.8) | 7170 (45.8) | 9730 (35.3) | 7690 (39.1) | 11100 (24.5) | 10800 (30.4)

6. Secondary Outcome: Cmax (Maximum Measured Concentration of the Ida in Plasma)
Description: Cmax. PK/PD sampling time: (p=predose, D=day)
  1. single medium or high dose, HS mid-age (45-64 yrs): D4: 8:55p, 9:00,9:10,9:30,10:00,11:00,13:00,15:00,19:00,21:00,01:00; D5: 9:00p, 21:00. D6: 9:00.
  2. single low or high dose, healthy elderly or mild RI: D4: 8:55p, 9:00,9:10,9:30,10:00,11:00,13:00,15:00,19:00,21:00,01:00; D5: 9:00; D6: 9:00; D7: 9:00; additional sampling for RI: D8: 9:00;D9: 9:00.
  3. high 2 doses, moderate RI: D4: 8:55p, 9:00, 9:10,9:30,9:55p, 10:00,10:10,10:30,11:00, 13:00, 15:00, 19:00, 21:00, 01:00; D5: 9:00; D6: 9:00; D7: 9:00; additional sampling for RI: D8:9:00; D9:9:00.
Time Frame: From Ida administration to 4 days post dose (details in description)
Population: PKS-Ida
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Groups:
- 220 mg/2.5 g HS 45-64 Years: HS mid-age (45-64 yrs) with dabigatran (DE) 220 mg/Ida 2.5g.
- 150 mg/1 g Mild RI (CL 60-90): Mild RI (CL 60-90) with dabigatran (DE) 150 mg/Ida 1g
Arm/Group | 220 mg/2.5 g HS 45-64 Years | 220 mg/2.5 g HS 45-64 Yrs Re-exposure | 220 mg/5 g HS 45-64 Yrs | 220 mg/1 g HS 65-80 Yrs | 220 mg/5 g HS 65-80 Yrs | 150 mg/1 g Mild RI (CL 60-90) | 150 mg/5 g Mild RI (CL 60-90) | 150 mg /2*2.5 g Moderate RI (CL 30-60)
Number analyzed (Participants) | 6 | 6 | 6 | 8 | 8 | 6 | 6 | 6
nmol/L | 15700 (14.3) | 14900 (12.0) | 25000 (16.9) | 5790 (16.4) | 28300 (28.9) | 6940 (19.4) | 32100 (17.4) | 25600 (11.6)

7. Secondary Outcome: Ae0-6 (Amount of Ida Eliminated in Urine From the Time Point 0 to Time Point 6 h)
Description: Ae0-6 (Amount of Ida Eliminated in Urine From the Time Point 0 to Time point 6 h).
  PK Urine sampling time:
  Urine sampling relative to DE administration: Planned times 72:00 - 73:55h, 73:55 - 80:00h, 80:00 - 86:00h, 86:00 - 98:00h, 98:00 - 122:00h, 122:00 - 146:00h; additional sampling for renal impaired: 146:00 - 170:00; 170:00 - 194:00h.
Time Frame: from 0 to 6 hours of post Ida dose (details in description)
Population: PKS-Ida: The PKS-Ida included all treated subjects who have received at least 1 dose of idarucizumab and who provided data for at least 1 secondary or other PK endpoint in any treatment period, which was judged as evaluable for PK and was not affected by (important) protocol violations relevant to the statistical evaluation of PK endpoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: umol
Arm/Group | 220 mg/2.5 g HS 45-64 Years | 220 mg/2.5 g HS 45-64 Yrs Re-exposure | 220 mg/5 g HS 45-64 Yrs | 220 mg/1 g HS 65-80 Yrs | 220 mg/5 g HS 65-80 Yrs | 150 mg/1 g Mild RI (CL 60-90) | 150 mg/5 g Mild RI (CL 60-90) | 150 mg /2*2.5 g Moderate RI (CL 30-60)
Number analyzed (Participants) | 6 | 0 | 6 | 8 | 8 | 6 | 6 | 6
umol | 13.5 (32.6) |  | 33.5 (60.0) | 1.97 (69.0) | 41.6 (13.7) | 2.60 (46.7) | 33.4 (48.9) | 31.3 (89.0)

ADVERSE EVENTS:
Time Frame: From the study drug administration up to start of follow-up period (from Day 1 to Day 35).
Groups:
- Dabigatran Etexilate (DE): subjects with Dabigatran etexilate (DE) treatment
- Low (1g) Idarucizumab Dose: Subjects with low 1g idarucizumab dose treatment
- Medium (2.5g) Idarucizumab Dose: Subjects with medium (2.5g) idarucizumab dose treatment
- High (5g) Idarucizumab Dose: Subjects with high (5g) idarucizumab dose treatment
- Low (1g) Placebo Dose: Subjects with low (1g) placebo dose treatment
- Medium (2.5g) Placebo Dose: Subjects with medium (2.5g) placebo dose treatment
- High (5g) Placebo Dose: Subjects with high (5g) placebo dose treatment
Arm/Group | Dabigatran Etexilate (DE) | Low (1g) Idarucizumab Dose | Medium (2.5g) Idarucizumab Dose | High (5g) Idarucizumab Dose | Low (1g) Placebo Dose | Medium (2.5g) Placebo Dose | High (5g) Placebo Dose
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/14 | 0/12 | 0/26 | 0/14 | 0/12 | 0/26
Other Adverse Events (participants affected / at risk) | 13/46 | 4/14 | 1/12 | 2/26 | 3/14 | 3/12 | 0/26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dabigatran Etexilate (DE) (N=46) | Low (1g) Idarucizumab Dose (N=14) | Medium (2.5g) Idarucizumab Dose (N=12) | High (5g) Idarucizumab Dose (N=26) | Low (1g) Placebo Dose (N=14) | Medium (2.5g) Placebo Dose (N=12) | High (5g) Placebo Dose (N=26)
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 7 | 3 | 1 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 4 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Application site dermatitis (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.